CLINICAL TRIAL: NCT06971926
Title: Improving the Early Childhood Social Assistance National Program PI-SUAS/Criança Feliz: Impact Evaluation of the Home Visits
Brief Title: PI-SUAS - Impact Evaluation of Home Visits
Acronym: PI-SUAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Grand Challenges Canada (Other); Fundação Maria Cecília Souto Vidigal (Unknown)
Responsible Party: Principal Investigator, Alexandra Brentani, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: TTS-2024-71139
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: early child development; home visit programs; impact evaluation; parenting practices

STUDY DESIGN:
Intervention Model Description: The intervention will be delivered to 50% of the participants during year 1. The rest will remain as a control group during year 1 and will receive the intervention after endline data collection
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Eligible children who will not receive the intervention (home-visits) during the study period
- Home visit group (Experimental): Home visit to improve parenting practives and child development
  Interventions: Behavioral: Home visist

INTERVENTIONS:
Behavioral: Home visist — Caregivers and children will receive home visits twice a month delivered by the social assistance service within the PI-SUAS/CF during 12 months
  Other Names: PI-SUAS Home visits
  Arms: Home visit group

SUMMARY:
Background: Early childhood, particularly from 0-36 months, represents a critical period of human development marked by rapid growth and skill acquisition. The brain undergoes accelerated development and is highly receptive to stimuli and experiences, which leave lasting marks and influence the individual's future. A nurturing environment-characterized by sensitivity to the child's health and nutritional needs, caregiver responsiveness, and emotional support-is especially vital in early childhood, in this period. Such an environment safeguards the child and their development from the detrimental effects of adverse socioeconomic conditions. Among early childhood development (ECD) programs, home visits have proven to be an effective strategy for promoting positive parenting and fostering child development, supported by long-term evidence.

Objective: This study aims to assess the impact of the enhanced methodology of the Primeira Infância no SUAS/Programa Criança Feliz (PI-SUAS/CF) on early childhood development outcomes through a randomized controlled trial (RCT).

Methods: A randomized controlled trial will be conducted across 6 municipalities in Brazil, focusing on vulnerable populations. Participants will include eligible families with children aged 18-20 months who are not yet enrolled in the program. Participants will be randomly assigned to either the intervention or control group. The intervention group will receive home visits based on the revised PI-SUAS/CF methodology, which emphasizes age- and culturally appropriate practices, caregiver responsiveness, and emotional support for 12 months. The control group will receive standard social assistance services without the enhanced home-visiting methodology. Primary outcomes will include cognitive, language, and socio-emotional development, assessed using validated tools. Secondary outcomes will focus on the quality of caregiver-child interactions and parental practices. Data will be collected at baseline and endline.

Results: It is hypothesized that the revised methodology will lead to significant improvements in child development outcomes compared to the control group. The flexible, adaptable approach is expected to enhance the quality and effectiveness of home visits across diverse contexts.

Conclusion: This trial will provide robust evidence on the effectiveness of an improved home-visiting methodology in promoting early childhood development among vulnerable populations. The findings will inform policy decisions and support the scaling of early childhood interventions globally.

DETAILED DESCRIPTION:
Early childhood, the period from conception to six years of age, is a crucial phase of human development, marked by rapid growth and skills acquisition. The brain undergoes accelerated development and is highly receptive to stimuli and experiences, which leave lasting impressions and influence the individual's future.

The early years of the 21st century have been marked by a large body of scientific evidence on child development, demonstrating that the environment induces epigenetic, immunological, and psychosocial adaptations. These adaptations begin with conception and produce lifelong effects. In other words, factors such as the quality of the physical and social environment in which the child lives; access to healthcare; interaction and engagement from caregivers; cognitive and emotional stimulation; proper nutrition; and exposure to chronic toxic stress and adversity have a profound and lasting impact on the child's life and future.

Brain plasticity refers to the central nervous system's ability to reorganize itself in response to external stimuli, through the development of new synapses, changes in gene expression, among other processes. Studies have shown that this ability is greatest early in life and declines over time. In addition to the concept of brain plasticity, science has established that complex skills are built upon fundamental ones. Thus, a child's development is a process of maturation and interaction with the environment, resulting in sequential progression of perceptual, motor, cognitive, language, socioemotional, and self-regulation skills.

All this evidence reinforces the importance of ensuring a healthy start to life and protecting children from harmful and detrimental factors to their development. While this period of life is filled with opportunities for learning and growth, it is also a time of great vulnerability to the effects of adversity.

A nurturing environment-characterized by a home setting that is attentive to the child's health and nutritional needs, caregiver responsiveness, and emotional support during early childhood, especially in the first two years of life-protects the child and their development from the damaging effects associated with poor socioeconomic conditions. Failing to provide such conditions and stimuli results in impaired full development of the child, with serious individual consequences such as chronic diseases in adulthood, lower academic achievement, and reduced labor market participation and income throughout adult life. On a societal level, the consequences include increased public health costs, the persistence and worsening of social inequality, and the loss of human capital.

Alongside the growing body of evidence, the discussion around the urgent need for policies and social programs to change the life trajectory of children in vulnerable social contexts has intensified. Typically, investments in the pediatric age group focus on the education of children over 7 years old and adolescents, leaving early childhood underserved by public policies and social programs. These findings justify investing in early childhood, yet they still do not fully answer which interventions are most effective in changing the developmental trajectory of the over 200 million children under the age of five, most of whom live in low- and middle-income countries-who do not reach their full potential.

Given that a nurturing early childhood environment is the primary essential determinant of human capital development followed by a high-quality education system, public programs and policies that support families and parents in creating such an environment are key to promoting healthy child development. Examples of such initiatives include paid maternity and paternity leave, support for breastfeeding in the workplace, the provision of quality childcare services, and access to free education. Among the interventions and policies focused on early childhood, more specifically, a key category stands out: programs that provide support and education for parents and caregivers to help them create a nurturing environment. Such an environment can break the intergenerational cycle of poverty, reduce social conflict, and mitigate other forms of stress. These programs share the common goal of modifying behaviors, increasing the frequency of positive interactions between caregivers and children, and strengthening their bond, thereby creating opportunities for learning. Several formats for these programs have been proposed and studied, among which home visits are particularly notable as an effective strategy for promoting positive parenting and, consequently, healthy child development, with long-term evidence supporting their benefits. As a result, numerous programs have been implemented globally. There is a broad consensus in the literature on the importance of early experiences for development and the effectiveness of early stimulation programs-especially through home visits-as a strategy with far-reaching results. However, to ensure that children and their families truly benefit from home visiting programs, attention must be paid to their implementation and quality. Access alone is not enough to improve outcomes for children and families. Several factors are essential, such as:

* the home visitor's understanding of the program and of child development;
* the bond they build with families;
* the suitability of the proposed activities and play for the child's age and context;
* sensitivity to local cultural specificities and the ability to tailor the service to individual needs;
* the supervision process, including ongoing support and training for the visitor;
* and fidelity to program content, among others. Nonetheless, achieving sustainable and high-quality results at scale has proven to be a major challenge, often resulting in a reduced impact of these programs on child development. Another obstacle has been the adaptation of interventions to diverse contexts and cultures, which has hindered the adoption and effectiveness of many programs.

The Criança Feliz Program / Early Childhood in SUAS In light of the global strategy for promoting child development, scientific evidence, and, at the national level, the approval of the Legal Framework for Early Childhood, which establishes the prioritization of actions for children aged 0-6, the Criança Feliz Program / Early Childhood in SUAS was established through Decree No. 8,869, of October 5, 2016 (later amended by Decree No. 9,579, of November 22, 2018). The program was created with an intersectoral approach and the goal of promoting the holistic development of children in early childhood, considering their family and life context. The Criança Feliz / Early Childhood in SUAS program (PCF) is a national initiative focused on promoting parenting and child development and is one of the largest home visiting programs in the world. The target population includes families with pregnant women and young children in socially vulnerable conditions. The program operates in a decentralized manner, being implemented at the municipal level with support from state and federal governments.

The PCF is based on two interconnected activities: home visits-which are the core component of the program-and intersectoral initiatives. For example, home visits are family-centered and respect diverse family arrangements; they aim to strengthen the bonds between children and their caregivers and empower those caregivers. At the same time, home visitors act as an extension of the social protection network. Being in close contact with socially vulnerable families, they can refer families to other public social services when needed.

The program's governance model is built on decentralized and integrated actions, promoting shared responsibility among various levels of government. Eligibility to participate in the PCF extends to states, municipalities, and the Federal District, provided they meet specific inclusion criteria.

Brazil is geographically divided into five regions, which are further divided into 26 states plus the Federal District, totaling 5,570 municipalities. In a proposal to reorganize the program based on data from May 2023, 75% (4,153) of these municipalities met the inclusion criteria for the Criança Feliz / Early Childhood in SUAS program. These criteria include having a Social Assistance Reference Center (CRAS), being registered in the national social service information system (CAD-SUAS) and having a minimum of 140 potential beneficiaries. Municipal participation varies by state-for example, Ceará and Roraima have 100% of eligible municipalities enrolled in the program, while Santa Catarina, Paraná, and Espírito Santo have fewer than 20% of their eligible municipalities actively participating.

Evaluations of the Early Childhood in SUAS / Criança Feliz Program The evaluations conducted on the program, including a randomized controlled trial designed to assess its implementation and impact across 30 Brazilian municipalities, have consistently pointed to the need for strengthening its implementation.

Among these evaluations, the impact and implementation assessment initiated in 2018 by the Federal University of Pelotas, both the Intention-to-Treat (ITT) and Local Average Treatment Effect (LATE) analyses found no significant evidence of differences between the intervention and control groups in terms of child development, responsive caregiving, disciplinary methods, or psychological attributes. The study revealed several implementation challenges, including inadequate coverage and deficiencies in the quality of home visits. Many of the observed visits lacked predefined content and did not take the child's age into account.

3. The Reorganization of the Early Childhood in SUAS / Criança Feliz Program In 2023, in response to the findings from various evaluations of the program and with the goal of strengthening it, a Technical Committee was established within the Tripartite Intermanager Commission (CIT) to implement the reorganization of the Criança Feliz / Early Childhood in SUAS program aiming to integrate the program into the Social Assistance Services and improving the quality of the visits.

4. Project to Improve the PI-SUAS/CF Program

In light of the need to enhance the Program, the project "Improvement of the PI-SUAS/CF Methodology" was launched in December 2023. The main innovation of the project, which was thoroughly discussed and approved by the federal government, is to propose the improvement of the home visit methodology to support Criança Feliz (PCF) home visitors in conducting visits for vulnerable populations throughout Brazil during pregnancy and the first three years of a child's life. This aims to contribute to achieving the overarching goal defined in the process mapping:

"To promote comprehensive early childhood development by strengthening social protection in the territory for children aged 0-6, caregivers, pregnant women, and families in situations of vulnerability, thereby contributing to reducing social inequalities." Based on this goal, and considering the weaknesses identified in previous impact evaluations, a revision of the visit content and staff training was carried out. The revised methodology was designed to be flexible and adaptable, aiming to improve visit quality in terms of age and cultural appropriateness.

Impact Evaluation Methodology Since the goal is to offer an impactful home-visit methodology to be used by all municipalities in Brazil (for the benefits to be directly measurable in tangible outcomes such as changes in parenting practices and the promotion of comprehensive child development), we will conduct an impact evaluation of the methodological revision.

ELIGIBILITY:
Inclusion Criteria: children enrolled in the social assistance vulnerability datasystem (CADUNico or Bolsa Família Recipient)

-

Exclusion Criteria:

* Children who receive or received home-visits from the social assistance PI-SUAS/CF

Ages: 18 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall child development | Age 2 - 3 years in after 12 months of intervention
  Children's overall development will be assessed using the Caregiver Reported Child Development Index - Credi Long form overall score. The scale ranges from 0 to 100, where a higher score indicates a child's development is progressing more positively. However, CREDI. Z-scores will be used to calculate and interpret the effect sizes.

SECONDARY OUTCOMES:
Parenting practices | Assessment after 12 months of intervention
  Parenting practices will be assessed using the Parenting and Family Adjustment Scales (PAFAS). The scores range from 0-42 points and higher overall PAFAS scores are interpreted as indicating greater levels of dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Brentani - Principal Investigator, PhD, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No